CLINICAL TRIAL: NCT03750175
Title: OPTImal PALliative Anti-epidermal Growth Factor Receptor Treatment in Metastatic Colorectal Cancer - Feasibility Study Investigating Circulating Tumor DNA for Treatment Decisions
Brief Title: OPTImal PALliative Anti-epidermal Growth Factor Receptor Treatment in Metastatic Colorectal Cancer -
Acronym: OPTIPAL-II
Status: Completed | Type: Observational
Sponsor: Karen-Lise Garm Spindler (Other)
Responsible Party: Sponsor-Investigator, Karen-Lise Garm Spindler, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: KFE1713
Record Dates: First submitted 2018-09-27; First posted 2018-11-21 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer Metastatic; Circulating Tumor DNA; KRAS Gene Mutation; NRAS Gene Mutation; BRAF Gene Mutation; Epidermal Growth Factor Receptor Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samles for circulating DNA analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Clinical utility of ctDNA analysis for treatment decision
  Use of ctDNA for KRAS, NRAS and BRAF testing prior to potential anti-EGFR monoclonal antibody treatment for metastatic colorectal cancer
  Interventions: Other: Plasma circulating DNA analysis

INTERVENTIONS:
Other: Plasma circulating DNA analysis — Clinical utility of ctDNA analysis for treatment decision

SUMMARY:
The present study will investigate the feasibility and clinical value of using circulating tumor DNA as selection for anti-epidermal growth factor receptor treatment for metastatic colorectal cancer.

DETAILED DESCRIPTION:
The primary aim of this prospective study is to investigate if cfDNA in plasma is feasible and reliable for selection of mCRC patients who will benefit of anti-EGFR monoclonal antibody therapy

Secondary, to analyze developments in mutational status as reflected by cfDNA in plasma during therapy and at time of progression

ELIGIBILITY:
Inclusion criteria

* Histopathologically verified metastatic colorectal cancer
* Indication for systemic palliative treatment with standard Anti-EGFR monoclonal antibodies
* Fit for therapy with EGFR inhibition
* Consent to treatment and sampling
* Measureable disease according to RECIST v 1.1
* Age ≥ 18

Exclusion criteria

* PS > 2
* Significant other cancer disease within 5 years of inclusion
* Conditions precluding sampling during therapy and treatment breaks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer and indication for palliative chemotherapy with potential anti-EGFR monoclonal antibody.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of ctDNA analysis for RAS mutation analysis | maximum 7 days
  Feasibility measures
  Identification of wildtype or mutated status and results delivered to clinicians
  * Initial clinical test results i.e. ctDNA mutations or wildtype status within 7 days
  * Detailed mutation type characterization is provided retrospectively.
  Failure parameters
  * Quality of samples; PB > 5%, CPP1 major loss < 10%
  * Transportation > 3 week days
  * Analysis > 3 working days
  * Total results delivered > 7 days.

SECONDARY OUTCOMES:
Retrospective concordance analysis | By end of study, expected after 3 years
  Retrospective comparison of tumor mutation and plasma mutation analysis at baseline
Disease control rate | 1 year
  Rate of disease control
OS | 3 years
  Overall survival rate
Resistance mutations | At time of progression, data analysis expected after 3 years
  Rate of Ectoderm mutations at time of progression
Lead time | At time of progression, data analysis expected after 3 years
  Calcualted lead time between radiologically detected progression and molecular biologically detected ( by Ectoderm and other resistance mutations) in the ctDNA.

CONTACTS AND LOCATIONS:
Overall Officials: Karen-Lise G Spindler, Study Chair — Department of Oncology, AUH, Dk
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Callesen LB, Sorensen BS, Pallisgaard N, Laugesen IG, Boysen AK, Spindler KG. Total cell-free DNA measurement in metastatic colorectal cancer with a fast and easy direct fluorescent assay. Mol Clin Oncol. 2022 Mar;16(3):64. doi: 10.3892/mco.2022.2497. Epub 2022 Jan 17. PMID 35154704